CLINICAL TRIAL: NCT05861323
Title: Feasibility of the Comfort Measures Only Time Out (CMOT) to Reduce Distress During Palliative Withdrawal of Mechanical Ventilation
Brief Title: Feasibility of the Comfort Measures Only Time Out (CMOT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Corey R. Fehnel, Division Chief, Neurocritical Care and Hospital Neurology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023P000160; K23AG066929 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-05-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: End of Life; Respiratory Failure; Ventilatory Failure; Coma; Aging
MeSH Terms: conditions — Death; Respiratory Insufficiency; Hypoventilation; Coma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Check-list Arm (Experimental): This feasibility study will test an ICU team-based time and and check-list intervention, the Comfort Measures Only Time Out (CMOT). The CMOT is designed to improve ICU team communication and better address patient comfort at the end of life. Participants in the CMOT are intensive care unit clinicians who are caring for a patient who is about to undergo palliative withdrawal of mechanical ventilation at the end of life. Feasibility will be assessed by: recruitment rates, protocol adherence, and acceptability to clinicians. Patient level outcomes such as distressful episodes/person-time alive will also be collected as a component of routine care in this exploratory analysis. The maximum time any participant (ICU clinician or patient) will be participating in the study is about four hours.
  Interventions: Behavioral: Comfort Measures Only Time out (CMOT)

INTERVENTIONS:
Behavioral: Comfort Measures Only Time out (CMOT) — This is a brief intensive care unit team (nurse, physician, advanced practice provider, respiratory therapist) intervention to improve communication and care of patients at end of life in the intensive care unit setting.
  Other Names: CMOT

SUMMARY:
Nearly 25% of Americans die in intensive care units (ICUs). Most deaths in ICUs are expected and involve the removal of ventilator support, or palliative withdrawal of mechanical ventilation (WMV). Prior work by the Principal Investigator (PI) found that patient suffering can be common; with 30-59% of patients going through this process experiencing distress. Thus, experts and national organizations have called for evidence to inform guidelines for WMV. This research study will 1) develop and refine a Comfort Measures Only Time out (CMOT) intervention consisting of a structured time out with check-list protocol for the ICU team (nurse, physician, respiratory therapist) to improve the process of WMV. and 2) Pilot test the CMOT intervention in 4 ICUs (2 medical/2 surgical) among 40 WMV patients.

DETAILED DESCRIPTION:
This study will field test an ICU team-based timeout and checklist intervention, the Comfort Measures Only Time Out (CMOT), in 6 cases with 2 ICU teams (3 cases/team) and then further refine based on ICU team and expert feedback to create a final version of the CMOT. Then pilot testing of the final CMOT intervention will occur in 4 ICUs (2 medical/2 surgical) among 40 WMV patients (20/ICU sub-type). There are two groups of human subjects for this study: 1) Patients (n=46)- eligibility criteria are: 1. age ≥ 18, 2. decision made for WMV by extubation (but not yet extubated). and 2) ICU clinicians (n= approximately 138) (ICU nurses, physicians/APPs, and respiratory therapists)- eligibility will include: 1. Age > 18, and 2. provision of direct care to the patient for at least 1-hour pre-extubation. Verbal consent will be obtained from ICU clinicians by the RA. During the preparation period, the research team will conduct seminars to inform the ICU team about the study recruitment and data collection procedures. Each morning during the 12-month recruitment period, a research assistant (RA) will ask the ICU team to identify potentially eligible patients.

Study Procedures:

Pilot-testing of the CMOT will be in 4 ICUs (2 medical/2 surgical) among 40 WMV patients (20 patients/ICU type). Feasibility will be assessed by: recruitment, protocol adherence, acceptability to providers (e.g. helpfulness, endorse future use), and outcome measurement: rates of distressful episodes/person time alive (primary outcome). Outcomes will be compared with OBSERVE-WMV historical controls to help inform the design of a larger trial.

ICU sites: The CMOT intervention will be delivered at the ICU team level in 2 medical ICUs (16 beds), and 2 surgical ICUs at BIDMC (22 beds). Each ICU will have a designated CMOT champion.

ICU provider training:

The RA will collaborate with the CMOT Champion to compile a list of 'targeted' providers for training including ICU nurses, physicians, residents/fellows, mid-level providers, and respiratory therapists expected to provide care in the ICU over the next 13 months. The list will be refreshed every 2 months to reach new staff. The goal will be to have all targeted providers complete either the in-person or online training seminar (see below) within one month from the initial start-up for "prevalent" providers, or from start time in the ICU for new providers. The RA will track provider participation based on seminar sign-in logs or online training completion (see below). Weekly reminders will be emailed to non-compliant providers. It is estimated there will be ~50-60 targeted providers per ICU (20-25 nurses, 10-15 physicians, 10-15 fellows/resident physicians/mid-level providers, and 5 respiratory therapists). Provider involvement will be voluntary with verbal informed consent obtained during orientation.

ELIGIBILITY:
Patient Inclusion Criteria

* Age ≥ 18
* Decision made for withdrawal of mechanical ventilation (WMV) by patient/surrogate and ICU team
* WMV has not yet occurred

Patient Exclusion Criteria

• None

ICU Clinician Inclusion Criteria:

* ICU nurse, Physician/Advance Practice Provider, or respiratory therapist
* Age ≥ 18
* Providing direct care to WMV patient for at least 1-hour pre-extubation

ICU Clinician Exclusion criteria:

• Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Study recruitment rate | At time of study completion (approximately 1-year)
  Recruitment rate will be determined by the number of eligible participants enrolled divided by the total number of eligible participants.
Protocol adherence | At time of study completion (approximately 1-year)
  Protocol adherence will be measured by the rate of completed CMOT check-lists among enrolled participants. This measure will be calculated as: the number of ICU clinician participants completing CMOT checklist divided by the number enrolled ICU clinician study participants.

SECONDARY OUTCOMES:
Recommendation for future use | Surveys will be completed at three hours of withdrawal of mechanical ventilation, or within 72-hours. The measure will be reported at time of study completion (approximately 1-year)
  Intensive care unit clinicians will complete a brief survey of their experience with the CMOT. The outcome measure will record whether the clinician would "recommend the CMOT be used in the future?" Response options will be recorded in the following categories: Yes, No, Don't Know, Prefer not to answer.

OTHER OUTCOMES:
Distressful episodes | Measurement will occur at the time of withdrawal of mechanical ventilation (WMV) and until death or three hours after WMV. The measure will be reported at time of study completion (approximately 1-year).
  The frequency of distressful episodes from the will be measured by trained intensive care unit nurses using the respiratory distress observation scale (RDOS) [Range 0-16, higher scores indicate greater distress] and clinical pain observation tool (CPOT) [Range 0-8, higher scores indicate greater pain]. A composite outcome measure of either RDOS more than 2 or CPOT > 0 will be used to define a distressful episode.

CONTACTS AND LOCATIONS:
Overall Officials: Corey R Fehnel, MD, MPH, Principal Investigator — Co-Director, Neuroscience Intensive Care Unit
Locations (1):
- Beth Israel Deaconess Medical center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer AG, Campbell ML, Hayes MM, Schwartzstein RM, White DB, Mitchell SL, Fehnel CR. Study protocol testing feasibility of the Comfort Measures Only Time out (CMOT) to reduce distress during palliative withdrawal of mechanical ventilation. Pilot Feasibility Stud. 2025 Aug 13;11(1):109. doi: 10.1186/s40814-025-01688-4. PMID 40804432